CLINICAL TRIAL: NCT06051890
Title: Assessing Optimal Extended-Release Buprenorphine (XRB) Initiation Points in Jail
Brief Title: Assessing Optimal XRB Initiation Points in Jail
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00926
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transition to Extended-Release Buprenorphine (XRB) (Experimental): Participants randomized to transition to treatment with XRB.
  Interventions: Drug: Extended-Release Buprenorphine (XRB)
- Sublingual Buprenorphine (SLB) Maintenance (Active Comparator): Participants randomized to remain on-treatment with SLB.
  Interventions: Drug: Sublingual Buprenorphine (SLB)

INTERVENTIONS:
Drug: Extended-Release Buprenorphine (XRB) — XRB (Sublocade) will be delivered as a pre-filled 2cc subcutaneous monthly injection, using a 300mg starting dose in most cases (100mg starting doses are available per the study team's clinical judgement). XRB consists of a depot injectable formulation in polymeric solution to the abdomen and releases buprenorphine over 28-days (4-weeks) by diffusion as the polymer biodegrades. Prior to an initial injection, the participant must be stable for several days or longer on sublingual buprenorphine (SLB) at doses of 8mg/day or higher. Participants will receive at least one XRB monthly injection prior to release, which investigators anticipate to usually be the 300mg dose. Some participants will be recruited earlier during the incarceration (or experience delayed release dates and then longer than anticipated incarcerations); XRB will be continued monthly from the time of induction to the day of release.
  Other Names: Sublocade
  Arms: Transition to Extended-Release Buprenorphine (XRB)
Drug: Sublingual Buprenorphine (SLB) — Maintenance of existing SLB prescription (treatment as usual).
  Arms: Sublingual Buprenorphine (SLB) Maintenance

SUMMARY:
This application describes a 3-year, randomized controlled trial. Eligible, consenting adults (N=200) with existing sublingual buprenorphine (SLB) prescriptions who enter Middlesex County House of Corrections (MCHOC) as pre-trial detainees will be randomized at admission on a 1:1 basis to be inducted onto extended-release buprenorphine (XRB) at the time of admission (experimental condition) or remain in SLB (E-TAU; all participants will also receive naloxone). The two approaches will be compared with regard to (1) the percentage of participants released from jail with at least 7 days of buprenorphine in their system, (2) percentage of participants continuing MOUD treatment in the community, and (3) infractions related to buprenorphine diversion.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated men able to provide written informed consent in English.*
* Unsentenced.
* Entering the facility with a prescription for SLB and receiving SLB for at least the previous 3 days.
* Minimum anticipated jail stay is 4 days.
* Willing to accept being randomized to the experimental condition (i.e., transitioning to XRB while incarcerated).

Exclusion Criteria:

* Sentenced.
* Allergy, hypersensitivity or medical contraindication to either medication.
* Chronic pain requiring opioid pain management or other contraindicated medications.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants released from jail with at least 7 days of buprenorphine in their system | Up to Month 6
  The percentage of participants leaving jail with at least 7 days of buprenorphine protection in their system. Measured using clinical and jail records.

SECONDARY OUTCOMES:
Percentage of participants continuing MOUD treatment in the community | Up to Month 9
  Percentage of participants who continue to access medication for opioid use disorder (MOUD) once released from jail. This will be based on community clinic records indicating admission and retention.

CONTACTS AND LOCATIONS:
Overall Officials: David Farabee, PhD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - Tufts University Health Sciences, Boston, Massachusetts
  - Baystate Health, Springfield, Massachusetts
  - Middlesex County House of Corrections, New Brunswick, New Jersey
  - NYU Langone Health - 180 Madison Ave, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the de-identified individual participant data collected during the trial will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: david.farabee@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to david.farabee@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.